CLINICAL TRIAL: NCT00004330
Title: Studies in Porphyria IV: Gonadotropin-Releasing Hormone (GnRH) Analogues for Prevention of Cyclic Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Purpose: Prevention
Other Study IDs: 199/11885; UTMB-445; UTMB-312
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Porphyria
Keywords: inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Porphyrias; Metabolism, Inborn Errors; Rare Diseases | interventions — Gonadotropin-Releasing Hormone

INTERVENTIONS:
Drug: luteinizing hormone-releasing factor

SUMMARY:
OBJECTIVES:

Assess whether chronic administration of gonadotropin-releasing hormone analogues is safe and effective for the prevention of cyclic attacks of acute porphyria in women.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: All patients receive a gonadotropin-releasing hormone (GnRH) analogue. Treatment begins on days 1 to 3 of a menstrual cycle.

Low-dose estrogen begins at approximately 3 months. All patients must have a daily calcium intake of at least 1 gram; supplements are allowed.

Patients are followed for at least 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Acute porphyria, i.e.: Acute intermittent porphyria Hereditary coproporphyria Variegate porphyria Definite cyclic attacks with severe abdominal pain and other porphyria symptoms during luteal phase of menstrual cycle only Attacks resolve completely within 5 days of onset of menses, i.e., no symptoms between attacks At least 4 to 6 attacks during the 6 months prior to entry More than half of these attacks must meet the following criteria: Readily distinguishable from menstrual cramps and premenstrual syndrome Required hospitalization for narcotic analgesics, phenothiazines, hematin, intravenous fluids, or other treatment Luteal attacks not requiring hospitalization must be similar in symptoms and differ only in severity No life-threatening porphyria attacks No cyclic abdominal pain unless caused by porphyria --Prior/Concurrent Therapy-- At least 6 months since ovulation suppression --Patient Characteristics-- Reproductive: Menstrual cycle 25-35 days for at least 6 months prior to entry Pelvic exam normal within 60 days prior to entry Pap smear normal, i.e., no dysplasia No amenorrhea No other menstrual abnormality No other gynecologic abnormality Negative pregnancy test Medically approved contraception required for 2 months prior to entry and throughout study OR at least 1 menstrual cycle following tubal ligation Other: No allergy to gonadotropin-releasing hormone analogues No clinically significant abnormal laboratory test results No medical contraindication to protocol treatment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1987-03

CONTACTS AND LOCATIONS:
Overall Officials: Karl E Anderson, Study Chair — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States